CLINICAL TRIAL: NCT05344976
Title: An Exploratory Clinical Study on the Safety and Efficacy of MSLN STAR-T Cells in Advanced Malignant Solid Tumors
Brief Title: MSLN STAR-T Cells in the Treatment of Advanced Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXYT-I-018
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSLN STAR-T cells (Experimental): The patients will receive one dose of MSLN STAR-T.The dosage ranges from1×10^7 to 1×10^8 STAR-T+/kg.
  Interventions: Biological: MSLN STAR-T cells

INTERVENTIONS:
Biological: MSLN STAR-T cells — Patients with advanced MSLN-positive solid tumors will be recruited, and autologous-derived MSLN-STAR-T cells will be infused intravenously at escalating doses of 1×10^7-1×10^8 MSLN-STAR-T cells. The CAR-T ratio will be monitored at predetermined times (day 0, day 4, day 7, day 10, day 14, day 28).

SUMMARY:
This is a single-center, single-arm, open-label Phase I study to evaluate the safety and efficacy of MSLN STAR-T cell immunotherapy in the treatment of advanced malignant solid tumors.

DETAILED DESCRIPTION:
This study is a single-center, dose-escalation, prospective, exploratory study to evaluate the safety and efficacy of MSLN STAR-T cells in patients with hepatocellular carcinoma. The study is divided into two phases: dose escalation and dose expansion. The total duration of each subject's participation in the study is expected to be 24 months, including the screening period, non-myeloablative chemotherapy pretreatment, cell infusion-observation period, and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old, ≤ 70 years old, gender is not limited;
2. Advanced malignant solid tumors confirmed by histology or cytology, including malignant mesothelioma (pleura, peritoneum, etc.), pancreatic cancer, ovarian cancer, intrahepatic bile duct cancer, lung cancer, gastric cancer, colorectal cancer, etc.;
3. Patients with advanced malignant solid tumors who have relapsed after systemic therapy, or who cannot tolerate existing therapy, including but not limited to:

   * Patients with malignant mesothelioma who have failed at least first-line therapy;
   * Patients with pancreatic cancer who have failed at least first-line therapy;
   * Patients with gastric cancer who have failed at least second-line therapy in the past;
   * Patients with ovarian cancer who have previously failed at least second-line platinum-sensitive or platinum-resistant therapy;
   * Patients with intrahepatic cholangiocarcinoma who have failed at least first-line therapy;
   * Patients with advanced non-small cell lung cancer (non-squamous cell carcinoma): positive for EGFR, ALK, ROS1, MET and other driver genes, disease progression or intolerance after targeted therapy; negative for EGFR, ALK, ROS1, MET and other driver genes If the subject has disease progression or intolerance after receiving ≥ 1 line of therapy in the past;
   * Patients with colorectal cancer who have failed at least second-line therapy.
4. Tumor tissue samples are positive for mesothelin (MSLN) (IHC test, positive rate > 10%);
5. There are measurable target lesions on imaging (according to RECIST1.1) at the time of screening, the long diameter of non-lymph node lesions is ≥1.0cm, or the short diameter of lymph node lesions is ≥1.5cm;
6. ECOG score 0-1 points;
7. Expected survival period ≥ 3 months;
8. Have the conditions to establish a peripheral blood mononuclear cell collection pathway, and have enough cells for STAR-T cell preparation;
9. Has good bone marrow and organ function:

   * Blood routine: absolute neutrophil count (ANC) ≥1.5×109/L; hemoglobin (Hb) ≥85g/L; platelet count ≥75×109/L;
   * Blood biochemistry: total bilirubin (TBIL) ≤ 2.5 times the upper limit of normal (ULN); aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 times the upper limit of normal (ULN) (for liver metastases) Patients may be ≤5 times ULN);
   * Serum creatinine (Cr) ≤ 1.5 times the upper limit of normal (ULN);
   * Coagulation function: International Normalized Ratio (INR), Activated Partial Thrombin Time (APTT) ≤1.5×ULN, patients with liver metastases should be ≤2×ULN;
   * Pulmonary function: with the lowest level of lung reserve, defined as CTCAE v5.0 ≤ grade 1 dyspnea and end-finger oxygen saturation ≥ 91% in the non-oxygen state.

Exclusion Criteria:

1. Those with uncontrolled active infection at the time of screening; those who meet one of the following:

   Hepatitis B surface antigen (HBsAg) positive and/or hepatitis B e antigen (HBeAg) positive, hepatitis B e antibody (HBe-Ab) and/or hepatitis B core antibody (HBc-Ab) positive and HBV-DNA copy number greater than the detection limit, hepatitis C antibody (HCV-Ab) positive and HCV-RNA copy number greater than the lower limit of detection, human immunodeficiency virus (HIV) antibody positive, Treponema pallidum (TP-Ab) antibody positive;
2. Patients with or with a history of central nervous system diseases, such as history of epilepsy, stroke, severe brain damage, aphasia, paralysis, etc.;
3. Patients with active brain metastases but who do not need any radiation, surgery or steroid therapy to control metastatic symptoms 1 month before screening can be enrolled;
4. Systemic lupus erythematosus, combined with active or uncontrolled autoimmune diseases (such as Crohns disease, rheumatoid arthritis, autoimmune hemolytic anemia, etc.);
5. Are receiving therapeutic dose or systemic glucocorticoid therapy (prednisone ≥ 20 mg/day or equivalent dose of other corticosteroids);
6. Toxicity or complications caused by previous interventions or treatments have not recovered to CTCAE v5.0 ≤ grade 2 or below (except for hair loss and abnormal values of laboratory tests judged by the investigator);
7. Previously received other genetically modified T cell products (such as MSLN CAR-T or TCR-T cells), or treatment targeting MSLN;
8. Patients who have received any of the following drugs or treatments within the specified time period prior to apheresis:

   * Received any chemotherapy within 2 weeks or 5 half-lives, whichever is shorter, prior to apheresis;
   * Received any macromolecule or small molecule targeted therapy such as monoclonal antibody, antibody-drug conjugate (ADC), double antibody, etc. within 4 weeks or 5 half-lives (whichever is shorter) before apheresis;
   * Received radiotherapy within 6 weeks before apheresis. If the disease progresses in the radiotherapy site, or there are CT and other image-positive lesions in other non-radiotherapy sites, the group is allowed to enter the group; if there are CT and other image-positive lesions in other non-radiotherapy sites, it is allowed to 2 weeks before harvest, radiotherapy is performed on a single lesion;
9. The presence of uncontrolled pleural effusion, pericardial effusion or ascites (ascites is defined as: ascites with positive signs of ascites on physical examination or ascites that needs to be controlled by intervention (only those with ascites shown by imaging without intervention can be included).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-04-14 (Estimated); Primary Completion 2024-10-14 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of adverse events | 3months
  Percentage of participants with adverse events.